CLINICAL TRIAL: NCT03204747
Title: Effect of Need to Void on Gait Speed in Multiple Sclerosis
Status: Completed | Type: Observational
Sponsor: Pierre and Marie Curie University (Other)
Responsible Party: Principal Investigator, Gérard Amarenco, Head of Neuro-urology department, Tenon hospital, Pierre and Marie Curie University
Other Study IDs: P GREEN 001
Record Dates: First submitted 2017-06-27; First posted 2017-07-02 (Actual); Last update posted 2019-07-19 (Actual); Status verified 2019-07

CONDITIONS: Multiple Sclerosis; Lower Urinary Tract Symptoms; Gait
Keywords: Gait speed; multiple sclerosis; lower urinary tract symptoms; overactive bladder
MeSH Terms: conditions — Multiple Sclerosis; Lower Urinary Tract Symptoms; Urinary Bladder, Overactive

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients enrolled: Patient with multiple sclerosis and lower urinary tract symptoms, age > 18, able to walk without human help on 50 meters, able to hold urine at least 3 minutes.
  A first record of gait will be at strong desire to void. A second record will be after void Gait records consist on : 3 10meter walk test and 1 Timed up and Go test.
  Interventions: Other: Observational study : gait speed

INTERVENTIONS:
Other: Observational study : gait speed — No intervention, only propose water and wait for need to void

SUMMARY:
Multiple sclerosis causes demyelinating lesions, which can induce multiple symptoms. If motor disorders are the most visible disability, urinary disorders are frequent, with prevalence from 32 to 86%. The first ones are due to pyramidal, cerebellar or proprioceptive lesions. The seconds are due to specific lesion in inhibitor/activator encephalic centers, or interruption on medullary conduction. It seems to be evident that walk and urinary disorders are link, because of similar anatomic ways and control process. Effect of bladder filling is well known on motoneuronal excitability. The effect of bladder filling on walk stay unknown, while medullary integration of these two functions is very close, in medullary cone.

Primary aim is to assess the effect of need to void on walk speed in multiple sclerosis with lower urinary tract symptoms. Secondary aim is to identify clinical or urodynamic factor link with major walk impairment when patients need to void.

Patient with multiple sclerosis over 18 years old, consulting for lower urinary tract symptoms in a tertiary center are included.

History and treatment, high, weigh, symptoms severity by USP score, cognitive impairment by MMSE score and last urodynamic data are recorded. Patient are asked to drink water until they feel a strong need to void, for which they would go to urinate at home.

Walk tests are realized in a specific place, with calm and no passage. A chair is placed at each end of the path. Toilets are just next to the hall where they realize the tests. A 10 Meters Walk Test is done during this condition, 3 times (only the intermediate 6 meters are recorded). They can take 30 seconds of rest between each try if necessary. One Timed up and go is done. Patient can use their habitual walking device. Speed walk asking is comfortable for the two test.

Next, patient can urinate. 3 post void residual volume with portable echography are done, and the higher is recorded.

Patient achieve the same walk tests after urinate, in the same order. They must use the same walking device.

Primary outcome is mean gait recorded for 10 meters walk test.

Secondary outcome is time for timed up and go test.

Individual variability between the 3 10MWT in the two conditions will be study.

Influence of age, EDSS, severity of symptoms, MMSE, detrusor overactivity on speed impairment will be study in secondary analysis.

ELIGIBILITY:
Inclusion Criteria:

* Multiple sclerosis
* Follow in neuro-urology for lower urinary tract symtpoms
* Able to walk 50 meters without human assistance
* able to hold on void during 3 minutes at least

Exclusion Criteria:

* actual urinary tract infection
* relapse in the last week
* Mini Mental State Examination < 10

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients consulting in a tertiary center in neuro-urology
Sampling Method: Non-Probability Sample
Enrollment: 71 (Actual)
Dates: Start 2017-02-27 (Actual); Primary Completion 2017-08-31 (Actual); Study Completion 2017-08-31 (Actual)

PRIMARY OUTCOMES:
Gait speed | 1 Day: at strong desire to void and just after void
  Gait speed calculated from 10 meter walk test. Only the 6 intermediate meters are recorded. Time is recorded by a manual chronometer. 3 records are done, mean time is calculated. Mean time is divided by 6 to obtain mean gait speed

SECONDARY OUTCOMES:
Time for Timed up and Go | 1 Day: at strong desire to void and just after void
  1 record is done for timed up and go test after a first training. Time is recorded by a manual chronometer
Variation of gait speed | 1 Day: for strong desire to void and post void
  Coefficient of variation is calculated from the 3 records of 10 meter walk test. It correspond to standard deviation/average.

CONTACTS AND LOCATIONS:
Overall Officials: Gérard Amarenco, PhD, Principal Investigator — GREEN GRC-01, Neuro-urology, hôpital Tenon
Locations (1):
- Service de Neuro-urology, hôpital Tenon, Paris, France